CLINICAL TRIAL: NCT02797223
Title: "Impacto de la Alopecia Inducida Por Quimioterapia en la Calidad de Vida de Mujeres Con cáncer de Mama"
Brief Title: "Impact of Chemotherapy-induced Alopecia on the Quality of Life of Women With Breast Cancer"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CAL-2016-20
Record Dates: First submitted 2016-05-27; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Chemotherapy-induced Alopecia
Keywords: alopecia; chemotherapy; breast cancer
MeSH Terms: conditions — Alopecia; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Semi-structured interviews — Qualitative phenomenological study. Data collection will be done through semi-structured interviews. Each interview will last between 60 and 90 minutes. It will be the same researcher who interviewed and analyze them.

SUMMARY:
The main objective of this qualitative phenomenological study is to understand the impact of chemotherapy-induced alopecia, the quality of life of women with breast cancer from this experience.

The study will be conducted in the day hospital oncology-hematology of the Hospital de la Santa Creu i Sant Pau. Data collection will be done through semi-structured interviews. About 12 to 14 interviews throughout the study was conducted. So in the study involved a total of between 12 and 14 women.

These will be recorded in voice and then transcribe and code. From reading and re-reading the patterns or data that relate to each other, thus establishing the categories (thematic analysis) were identified. These categories describe the experiences of the participants alopecia.

DETAILED DESCRIPTION:
The main objective of this study is to understand the impact of chemotherapy-induced alopecia, the quality of life of women with breast cancer from this experience.

Therefore, it is a qualitative phenomenological study. The problem of the study is the impact of alopecia as a side effect of chemotherapy in women with breast cancer in the areas of privacy, welfare, sexuality and femininity, self-esteem, social relations and the world of work.

The study will be conducted in the day hospital oncology-hematology of the Hospital de la Santa Creu i Sant Pau. Data collection will be done through semi-structured interviews. Each interview will last between 60 and 90 minutes will be the participant who decides the date and time. The site will be a day hospital office.

It will be the same researcher who interviewed and analyze them. To make the selection of participants with an opinion sampling is performed. Attracting participants who are patients in the study investigator.

Inclusion criteria are: being female, of age, suffer from breast cancer, receive or have received chemotherapy have the side effect of alopecia and alopecia file or have filed at the time of the interview. Excluded from the study participants to present cognitive impairment, intellectual disability, presence of disease that prevents the story of their experience and / or not be able to sign the study informed orally and written consent.

About 12 to 14 interviews throughout the study was conducted. So in the study involved a total of between 12 and 14 women.

These will be recorded in voice and then transcribe and code. From reading and re-reading the patterns or data that relate to each other, thus establishing the categories (thematic analysis) were identified. These categories describe the experiences of the participants alopecia.

In a first phase of the project only 6 interviews will be conducted, as it requires the presentation of preliminary results as part of a master work carried out by the principal investigator. Subsequently, the remaining interviews will be conducted and the results will be analyzed in its entirety.

These six interviews are conducted between June and July 2016 total planned month duration of the study: 8 months.

Ethical considerations of this study are that to participate in the study informed consent is required describing procedures and the role of the participants, stressing the voluntary and total freedom to leave when they want. where the information sheet explaining why the study, its purpose and the importance of their participation among others shall also be included.

In addition, interviews will be recorded only voice and difficult to identify the participants. Finally, compliance with current regulations concerning the confidentiality and anonymity of the data is guaranteed.

This study does not have sources of funding.

ELIGIBILITY:
Inclusion Criteria:

* Being female, > 18 years old, suffer from breast cancer, receive or have received chemotherapy have the side effect of alopecia and alopecia file or have filed at the time of the interview.

Exclusion Criteria:

* Participants to present cognitive impairment, intellectual disability, presence of disease that prevents the story of their experience and / or not be able to sign the study informed orally and written consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women suffered breast cancer and alopecia post treatment
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 8 months
  Impact of chemotherapy-induced alopecia on the quality of life of women with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jorgina Serra, Nurse, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided